CLINICAL TRIAL: NCT03500562
Title: Daclatasvir-Based Therapy Safety Surveillance in Chinese Patients With Chronic Hepatitis C
Brief Title: Study of Daclatasvir-based Therapy in Chinese Participants With Chronic Hepatitis C (CHC)
Status: Terminated | Type: Observational
Why Stopped: Insufficient Enrollment
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Other Study IDs: AI444-396
Record Dates: First submitted 2018-04-10; First posted 2018-04-18 (Actual); Last update posted 2021-09-01 (Actual); Status verified 2021-08

CONDITIONS: Chronic Hepatitis C
MeSH Terms: conditions — Hepatitis C, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- HCV participant population in China

SUMMARY:
Study is a non-interventional, prospective, multicenter post marketing surveillance study to determine the safety of daclatasvir based therapy

ELIGIBILITY:
Inclusion Criteria:

* Participants 18 years of age and older
* Participants with Chronic Hepatitis C virus (CHC) who are eligible for treatment with branded DCV-based therapy as indicated in the locally approved label

Exclusion Criteria:

* Participants under the age of 18

Other protocol defined inclusion/exclusion criteria could apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients who receive branded DCV-based therapy in the real-world treatment setting for the first time under the approved indications.
Sampling Method: Probability Sample
Enrollment: 3 (Actual)
Dates: Start 2018-05-08 (Actual); Primary Completion 2019-03-29 (Actual); Study Completion 2019-03-29 (Actual)

PRIMARY OUTCOMES:
Number of adverse events (AEs) | Approximately 72 weeks
Number of serious adverse events (SAEs) | Approximately 72 weeks

SECONDARY OUTCOMES:
Number of participants who discontinue therapy due to an AE | Approximately 72 weeks
Effectiveness of daclatasvir DCV-based therapy | Approximately 72 weeks
  As measured by Sustained virologic response 12 weeks after the end of treatment (SVR12) Achieved SVR12: Hepatitis C virus (HCV) RNA below the lower limit of quantification (LLOQ)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (2):
- China (2):
  - Local Institution, Beijing, Beijing Municipality
  - Local Institution, Guangzhou, Guangdong

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: Investigator Inquiry Form — https://www.bms.com/researchers-and-partners/investigator-inquiry-form.html
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm